CLINICAL TRIAL: NCT07306546
Title: Effectiveness of Hydrogen Water Intervention on Acute Oral Inflammation, Oral Microbiota, and Pain Following Free Flap Reconstruction in Patients With Oral Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20250332
Record Dates: First submitted 2025-12-07; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Oral Squamous Cell Carcinoma (OSCC); Postoperative Pain; Postoperative Oral Mucositis; Free Flap Reconstruction; Oral Cancer
Keywords: Hydrogen water; Oral cancer; Free flap reconstruction; Pain assessment; Salivary Biomarkers
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Pain, Postoperative; Mouth Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen Water Oral Care Group (Experimental): This study adopts a randomized controlled trial (RCT) design with an equal allocation pretest-posttest approach and double-blind methodology. Eligible patients who underwent microsurgical free flap reconstruction for oral cancer were enrolled once their postoperative condition stabilized. They were randomly assigned in a 1:1 ratio to the experimental group using a computer-generated randomization table. Immediately after allocation, the first saliva collection (T0) was performed. Participants in the experimental group received daily hydrogen water oral care, using hydrogen water with a concentration of 1.1 mg/L and a dissolution stability of at least 12 hours. A second saliva collection (T1) was conducted on Day 7 of the intervention to evaluate changes in salivary inflammatory biomarkers, oral microbiota, and pain.
  Interventions: Other: Hydrogen Water Oral Care
- Water Oral Care Group (Placebo Comparator): Patients assigned to the control group through the same computer-generated 1:1 randomization process received tap water oral care. The first saliva collection (T0) was completed immediately after group allocation. Participants in the control group performed oral care daily using tap water at time points and frequencies identical to those of the experimental group. The second saliva collection (T1) occurred on Day 7 of the intervention to compare the effects of different oral care solutions on changes in salivary inflammatory biomarkers, oral microbiota, and pain.
  Interventions: Other: Water Oral Care

INTERVENTIONS:
Other: Hydrogen Water Oral Care — The research team provided hydrogen water daily according to group assignment. The hydrogen water used in this study contained 1.1 mg/L of dissolved hydrogen with a stability of no less than 12 hours. Participants performed oral care using the hydrogen water following standardized instructions. Saliva samples were collected at T0 (immediately after randomization) and T1 (Day 7 of the intervention) to assess changes in inflammatory markers, oral microbial composition, and pain levels during the intervention period.
  Arms: Hydrogen Water Oral Care Group
Other: Water Oral Care — The research team provided tap water for oral care daily, following the same procedures, frequency, and schedule as the experimental group, but without the active hydrogen component. Saliva samples were collected at T0 (immediately after randomization) and T1 (Day 7 of the intervention) to establish a placebo-controlled comparison of outcomes related to inflammatory markers, microbial profiles, and pain.
  Arms: Water Oral Care Group

SUMMARY:
This study employs a Randomized Controlled Trial (RCT) design. Patients diagnosed with oral cancer by the attending physician and who meet the inclusion criteria will be admitted to the study after receiving a full explanation of the study objectives, intervention methods, potential risks, and participant rights from the research team upon their stable transfer to the plastic surgery ward post-operation. Written consent will be obtained from the patient and/or their legally authorized representative after adequate informed consent has been provided, before they are enrolled in the study.

DETAILED DESCRIPTION:
The study adopts a Randomized Controlled Trial (RCT) design. Patients diagnosed with oral cancer by the attending physician and who meet the inclusion criteria are enrolled in the study upon their stable transfer from the Intensive Care Unit (ICU) to the plastic surgery ward post-operation.

The research team will personally explain the study objectives, intervention methods, potential risks, and participant rights to the subjects (and/or their legally authorized representatives) and provide written documentation. After addressing all questions, informed consent is obtained, and the subject is enrolled in the study.

Subjects are then assigned via computer-generated randomization at a 1:1 ratio. The experimental group (18 individuals) receives hydrogen-rich water oral care. The hydrogen-rich water is delivered daily after its concentration is measured.

Oral integrity is assessed using the Oral Assessment Guide (OAG), which includes 6 items: lips, tongue, saliva, oral mucosa, gums, and teeth, scored from 1 to 3 points. The minimum score is 6, and the maximum score is 18.

Oral care frequency is based on the OAG score:

6-10 points: Oral care once per shift. 11-14 points: Oral care once every 4 hours. 15-18 points: Oral care once every 2 hours. Oral care involves using a sponge toothbrush dipped in hydrogen-rich water (concentration 1.1 mg/L) to gently brush the mucosa, maxilla/mandible (upper/lower jaws), and tongue. This is continuously performed for 7 days.

The control group (18 individuals) receives plain boiled water for oral care, with the same frequency as the experimental group. The research team will daily record the subjects' compliance and any adverse reactions.

During the intervention period, both groups receive identical postoperative care and health education in the plastic surgery ward.

The research team will collect the first sample (pre-test, T0) when the patient is transferred from the ICU to the plastic surgery ward, and the second sample on the 7th day post-operation (T1). Saliva samples will be collected at both time points to evaluate oral inflammatory markers (such as IL-1$\beta$, IL-6, IL-10, TNF-α) and the oral microbiome (analyzed by RT-PCR detection of the 16S rRNA gene sequence)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with oral cancer and receiving microsurgical free flap reconstruction.
* Age 18 years or older.
* Conscious and able to follow study instructions.
* Able to communicate without difficulty in Mandarin, Taiwanese, or through written communication.

Exclusion Criteria:

* Abnormal salivary gland function or severe xerostomia.
* Recent use of antibacterial mouthwash or antibiotic therapy that may affect oral microbiota.
* Presence of severe bacterial or viral oral infections, or significant periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
IL-1β、IL-6、IL-10、TNF-α | Baseline (T0) and Day 7 (T1)
  Salivary IL-1β、IL-6、IL-10、TNF-α concentration will be measured to assess the anti-inflammatory effect of hydrogen water oral care in postoperative oral cancer patients. Measurements will be used to evaluate changes in inflammation between baseline and Day 7.
Oral Assessment Guide (OAG) Score | Baseline (T0) and Day 7 (T1)
  Change in total OAG score from baseline to Day 7 will be used to evaluate oral mucosal integrity.

CONTACTS AND LOCATIONS:
Overall Officials: I-SHAN CHOU, MS, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital

IPD SHARING:
Plan to Share IPD: No